CLINICAL TRIAL: NCT06549829
Title: Nutrition-Optimized Prehabilitation's Impact on Perioperative Outcomes in Primary Hepatocellular Carcinoma: a Randomized Controlled Trial
Brief Title: The Effect of Nutrition-optimized Prehabilitation on Perioperative Intervention in Primary Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0344
Record Dates: First submitted 2024-05-13; First posted 2024-08-12 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutritional optimization-led triple prehabilitation Intervention (Experimental): Nutritional optimization-led triple prehabilitation
  Interventions: Other: Nutritional optimization-led triple prehabilitation Intervention
- Conventional triple prehabilitation Intervention (Other): Conventional triple prehabilitation
  Interventions: Other: Conventional triple prehabilitation Intervention

INTERVENTIONS:
Other: Nutritional optimization-led triple prehabilitation Intervention — The nutritional status of the patients was assessed together with the clinical nutritionist to develop an individualized nutritional plan. The experimental group used ordinary dietary supplementation + transoral nutritional supplementation, and the control group used ordinary dietary supplementation. The target energy was basal energy metabolism level * physical activity level, physical activity level was male: 1.55 female: 1.56; basal energy level was basal metabolism standardized value * body weight (basal metabolism standardized value for obese patients was 25; basal metabolism standardized value for normal or emaciated patients was 30). Add 600kcal capacity supplement to this. Exercise workouts focused on increasing lung capacity and cardiorespiratory tolerance. Specialized psychological interventions.
  Arms: Nutritional optimization-led triple prehabilitation Intervention
Other: Conventional triple prehabilitation Intervention — Conventional triple prehabilitation: ordinary dietary supplementation; exercise workouts focused on increasing lung capacity and cardiorespiratory tolerance; specialized psychological interventions.
  Arms: Conventional triple prehabilitation Intervention

SUMMARY:
The aim of this project is to investigate the effect of triple prehabilitation led by nutritional optimization in liver cancer patients' surgery. It improves the preoperative nutritional status of cancer patients, reduces the incidence of early postoperative complications, promotes postoperative recovery, and improves the quality of patients' survival. Patients were randomized into experimental and control groups based on exclusion and inclusion criteria. Nutritional interventions and exercise and psychological interventions for patients. Interventions will continue for two weeks prior to surgery. Routine clinical blood tests will be performed at the time of enrollment, on the first day before surgery and on the first, third and fifth days after surgery. Enrolled patients were followed up by telephone or outpatient clinic at 1,3,6 months postoperatively.

DETAILED DESCRIPTION:
Study subgroups: experimental group (nutritional optimization-led triple prehabilitation), control group (conventional triple prerehabilitation)

1. Enrollment Criteria

   ①Patients diagnosed with primary liver cancer.
   * Patients between 18 and 70 years old.

     * Patients who are feasible for surgical treatment after clinical evaluation. ④Major organ function meets the following conditions: neutrophil count >1.5*109/L /L; platelet count >100* 109/L; hemoglobin >90g/L; transaminase and creatinine <twice the upper limit.
2. Exclusion criteria

   * Patients with liver metastases or combined with other tumors. ② Patients with allergy to the ingredients of nutritional preparations.

     * Patients who cannot eat by mouth.

       * Patients with severe malnutrition that cannot be corrected by oral nutrition. ⑤ Patients with hyperthyroidism, fistula, and combined digestive system diseases.
3. Intervention measures The nutritional status of the patients was assessed together with the clinical nutritionist to develop an individualized nutritional plan. The experimental group used normal dietary supplementation + oral nutritional supplementation, and the control group used normal dietary supplementation. Target energy was defined as basal energy metabolism level*physical activity level, which was 1.55 for men and 1.56 for women; basal energy level was defined as basal metabolism standard value*body weight. Depending on the patient, a 20% increase in energy intake is calculated on top of the target energy. One scoop of oral nutritional powder has an energy of 27.5kcal, and the dose of nutritional powder needed is calculated from the increased energy intake value. The required amount of powder should be taken orally in 200ml of warm water three times a day, and the exact time of taking the powder should be customized according to the patient's condition.

   Other interventions:

   A personalized exercise program was developed with the rehabilitation physician, and the experimental and control groups underwent exercise to increase lung capacity and cardiorespiratory tolerance: respiratory exercise was included: the patients were guided to learn to cough and cough up sputum with deep breaths before the operation, and the respiratory trainer was used to carry out bedside training. The patients were instructed to learn to cough and cough up sputum with deep breaths before surgery. Exercise planning: aerobic exercise (jogging or walking) three times a day for 15 minutes.

   The experimental group and the control group underwent psychiatric intervention: patients were psychologically evaluated according to the Hospital Anxiety and Depression Scale (HADS), and the scores of the anxiety and depression subscales were as follows: 0-7 was negative; 8-10 was mild; 11-14 was moderate; and 15-21 was severe. Patients with anxiety tendencies were counseled at least three times during the preoperative week and given medication if necessary. At the same time, the patients were guided to self-psychological counseling: no less than 15 minutes before bedtime every day.At the same time, patients were guided to self-help psychological guidance: every day before bedtime, they should listen to soothing music for at least 15 minutes, which was provided by the project team.

   Intervention time: Nutritional, exercise and psychological interventions will continue for two weeks before surgery. Nutritional, exercise and psychological interventions will continue for two weeks before surgery.

   The patients will undergo routine clinical blood tests at the time of enrollment, 1 day before the operation and the 1st, 3rd and 5th days after the operation.
4. Follow-up The patients will be followed up by telephone or outpatient clinic at 1, 3, and 6 months after the operation; the patients' clinical data will be recorded.

The relevant clinical data during the process will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary liver cancer.

  * Patients between the ages of 18 and 70.

    * Patients who are feasible for surgical treatment after clinical evaluation. ④Major organ function meets the following conditions: neutrophil count >1.5*109/L; platelet count >100* 109/L; hemoglobin >90g/L; transaminase and creatinine <twice the upper limit.

Exclusion Criteria:

* Patients with liver metastases or combined with other tumors. ②Patients with allergy to the ingredients of nutritional preparations.

  * Patients with severe malnutrition who cannot eat by mouth. ④Patients with hyperthyroidism, fistula, and combined digestive system diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative serum prealbumin | One day after surgery, three days after surgery, five days after surgery
  peripheral blood
Postoperative transferrin | One day after surgery, three days after surgery, five days after surgery
  peripheral blood
Postoperative retinol-binding protein | One day after surgery, three days after surgery, five days after surgery
  peripheral blood

SECONDARY OUTCOMES:
Postoperative Six-minute walk test (6MWT) | One week after surgery
  walk test for six minutes
grading and incidence of various types of complications | one month after surgery
  complications grade and incidence
postoperative length of stay | stay hospital time, an average of 10 days
  stay hospital time
30-day readmission rate | postoperative for 30 days
  readmission rate
patient long-term quality of life indicators (6 months) | during postoperative for 6 month
  life quality

OTHER OUTCOMES:
Drainage tube removal time | Postoperative, an average of 3 days
  remove abdominal drainage

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Ding, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin Y, Zheng L, Fang K, Zheng Y, Wu J, Zheng M. Proportion of liver cancer cases and deaths attributable to potentially modifiable risk factors in China. Int J Epidemiol. 2023 Dec 25;52(6):1805-1814. doi: 10.1093/ije/dyad100. PMID 37431632
- [Background] Zhou YM, Zhang XF, Li B, Sui CJ, Yang JM. Postoperative complications affect early recurrence of hepatocellular carcinoma after curative resection. BMC Cancer. 2015 Oct 14;15:689. doi: 10.1186/s12885-015-1720-0. PMID 26466573
- [Background] Noba L, Rodgers S, Chandler C, Balfour A, Hariharan D, Yip VS. Enhanced Recovery After Surgery (ERAS) Reduces Hospital Costs and Improve Clinical Outcomes in Liver Surgery: a Systematic Review and Meta-Analysis. J Gastrointest Surg. 2020 Apr;24(4):918-932. doi: 10.1007/s11605-019-04499-0. Epub 2020 Jan 3. PMID 31900738
- [Background] Forsmo HM, Pfeffer F, Rasdal A, Sintonen H, Korner H, Erichsen C. Pre- and postoperative stoma education and guidance within an enhanced recovery after surgery (ERAS) programme reduces length of hospital stay in colorectal surgery. Int J Surg. 2016 Dec;36(Pt A):121-126. doi: 10.1016/j.ijsu.2016.10.031. Epub 2016 Oct 22. PMID 27780772
- [Background] Davis JF, van Rooijen SJ, Grimmett C, West MA, Campbell AM, Awasthi R, Slooter GD, Grocott MP, Carli F, Jack S. From Theory to Practice: An International Approach to Establishing Prehabilitation Programmes. Curr Anesthesiol Rep. 2022;12(1):129-137. doi: 10.1007/s40140-022-00516-2. Epub 2022 Feb 18. PMID 35194410